CLINICAL TRIAL: NCT04284891
Title: The Epidemiology of Critical Respiratory Diseases in Ex-preterm Infants Admitted to the Pediatric Intensive Care in Vietnam
Brief Title: Critical Respiratory Diseases in Ex-preterm Infants in PICU
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Phuc Huu Phan, Deputy Director of Pediatric Intensive Care Unit, National Children's Hospital, Vietnam
Other Study IDs: 2019-03
Record Dates: First submitted 2019-09-21; First posted 2020-02-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Infant, Premature, Diseases; Respiratory Disease; Respiratory Failure; Premature Birth
Keywords: Respiratory Diseases, ex-prematurity; Respiratory Failure; Pediatric Intensive Care
MeSH Terms: conditions — Infant, Premature, Diseases; Respiration Disorders; Respiratory Insufficiency; Premature Birth; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature birth is the leading cause of death in children younger than 5 years old worldwide, especially in low- and middle-income countries. Premature infants who survive are at greater risk of a range of short-term and long-term health consequences. Common long-term health morbidities among children who are born prematurely include cerebral palsy, infections (particularly respiratory infections), bronchopulmonary dysplasia, feeding difficulties, hypoxic-ischemic encephalopathy, visual and hearing problems. Re-hospitalization occurs frequently during first few years of life among ex-premature infants with respiratory illness. This leads to increased financial burden for health care system and families. The impact of prematurity on the health care system, especially on pediatric intensive care units (PICUs) has mainly been evaluated in high income countries. Little is known about long term health outcomes of ex-premature infants and their impact on the cost to health care system in low- and middle-income countries. This pilot, single institution, observational study aims to determine the prevalence, course of the diseases, and outcomes of ex-premature infants with respiratory illnesses who are admitted to a PICU of a tertiary children's hospital in Vietnam. Investigators will determine the epidemiology of respiratory illness, and the resource utilization for these children in the PICU. To achieve these aims, the investigators will prospectively screen and recruit all children aged less than 2 years old admitted to the PICU with respiratory illness/failure and collect pertinent clinical data. The study participants will be follow-up until PICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≤ 2 year olds with respiratory diseases admitted to pediatric intensive care unit of Vietnam National Children's Hospital

Exclusion Criteria:

* Nil

Ages: 30 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients aged ≤ 2 year olds with respiratory diseases
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of ex-premature infants aged < 2 years admitted to Pediatric Intensive Care Unit (PICU) | Through study completion, an average of 1 year
  The percentage of ex-premature patients to the total number of patients aged ≤ 2 years age admitted to PICU over a defined period
Percentage of ex- premature infants aged < 2 years admitted to PICU with critical respiratory diseases. | Through study completion, an average of 1 year
  The percentage of ex-premature patients to the total number of patients aged ≤ 2 years age with respiratory illness admitted to PICU over a defined period

SECONDARY OUTCOMES:
Percentage of identified pathogens of critical respiratory diseases among study participants | Up to 60 days
  Proportion of identified etiologies of critical respiratory diseases among participants will be reported
Number of participants with all-cause mortality | Up to 60 days
  The number of participants who died due to any cause while on the treatment will be assessed
Time from start to end of mechanical ventilation | Up to 60 days
  Time from start to end of mechanical ventilation will be measure
Time from pediatric intensive care unit (PICU) admission to PICU discharge | Up to 60 days
  The duration for how long the participant remained in the PICU that is the time from PICU admission to PICU discharge will be measured
Percentage of participants receiving mechanical ventilation support | Up to 60 days
  Percentage of participants receiving mechanical ventilation support will be reported. Mechanical ventilation support include invasive and non-invasive mechanical ventilation.
Percentage of participants receiving diagnostic imaging services | Up to 60 days
  Percentage of participants receiving diagnostic imaging services will be reported. Diagnostic imaging services include chest x-ray, chest computer tomography, cardiac ultrasound.
Percentage of participants receiving microbiological diagnostics | Up to 60 days
  Percentage of participants receiving microbiological diagnostics will be reported. Microbiological diagnostics include bacterial cultures and polymerase chain reaction (PCR) tests

CONTACTS AND LOCATIONS:
Overall Officials: Phuc H Phan, MD, Principal Investigator — Vietnam National Children's Hospital; Jan Hau Lee, MD, Principal Investigator — Duke-NUS Medical, Singapore
Locations (1):
- Vietnam National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No